CLINICAL TRIAL: NCT05501847
Title: Prevalence of Cardiac Amyloidosis in Patients With Hospitalization for Acute Heart Failure in the French West Indies
Brief Title: Heart Failure: Don't Forget the Role of Amyloidosis
Acronym: TEAM-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20_RIPH2-23
Record Dates: First submitted 2022-08-08; First posted 2022-08-16 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure
Keywords: Ventricular Hypertrophy; Amyloidosis Cardiac; Transthyretin gene mutation
MeSH Terms: conditions — Heart Failure; Amyloid Neuropathies, Familial

STUDY DESIGN:
Intervention Model Description: Prospective multicenter interventional study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with ventricular hypertrophy (No Intervention): Screening for cardiac amyloidosis in a patient with heart failure and ventricular hypertrophy is performed as part of routine care according to a standardised care protocol that follows the Gullimor algorithm.
- Patient with no ventricular hypertrophy (Experimental): In the context of TEAM-HF research, the heart failure patient without ventricular hypertrophy will undergo a bone scan.
  If the diagnosis of amyloidosis is most often suspected on the electrocardiogram and cardiac echography, only cardiac MRI or bone scan with diphosphonates (for transthyretin amyloidosis) can make the diagnosis.
  Interventions: Radiation: Patient with no ventricular hypertrophy

INTERVENTIONS:
Radiation: Patient with no ventricular hypertrophy — Patients without LVH ≥ 12 mm will routinely receive a bone scan as part of the study.
  In case of cardiac fixation on bone scan, the patient will be managed as part of routine care according to a standardized care protocol that follows Guillmor's algorithm: monoclonal abnormality testing on biological blood samples +/- genotyping, in order to specify the senile or mutated character of TTR cardiac amyloidosis and to give the genotype.
  Arms: Patient with no ventricular hypertrophy

SUMMARY:
Heart failure is defined as the inability of the heart to provide sufficient output to meet the needs of the body.

It can occur in the course of a myocardial infarction, angina pectoris, hypertension, etc. Its frequency increases with age.

It is a major public health problem.

Heart failure first appears during exercise, then at rest. Initially, the heart tries to adapt to the loss of its contraction force by accelerating its beats (increase in heart rate), then it increases in volume (thickening of the walls or dilation of the cardiac cavities). This extra workload for the heart eventually leads to heart failure.

Cardiac amyloidosis is a possible cause of the disease in the West Indian population.

Cardiac amyloidosis is a rare disease related to our own proteins that will accumulate and cluster together to form abnormal protein deposits that will eventually lead to heart failure.

Cardiac amyloidosis particularly affects West Indians, due to the high frequency in this population of a genetic anomaly associated with the disease: the Valine 122 Isoleucine (Val122l) mutation of the transthyretin gene (protein transthyretin in which isoleucine is substituted for valine at position 122 (Ile 122)).

Early detection of amyloidosis appears essential for the implementation of appropriate therapies and therefore for an improvement in patient survival.

For this it seems important to better specify the frequency of cardiac amyloidosis in heart failure in the French West Indies.

DETAILED DESCRIPTION:
The heart supplies the organs with oxygen and nutrient-rich blood. During exercise, the heart adapts by increasing the rate of contraction and the rate of blood flow.

Heart failure occurs when the heart loses its muscular strength and its normal capacity to contract; it no longer pumps enough blood to allow the organs to receive enough oxygen and nutrients, which are essential for their proper functioning.

This syndrome is frequent and serious with a prevalence of 2 to 3% in Europe and a high morbidity and mortality (1st cause of hospitalization with more than 150,000 hospitalizations per year in France, a mortality of 50% at 5 years, i.e. more than most cancers). This mortality is even higher in the West Indies, with an excess of premature mortality related to heart failure of +32.9% in Martinique and +86.9% in Guadeloupe compared with metropolitan France (average annual mortality rate for heart failure in 2008-2010 per 100,000 in habitants under 65 years of age).

Some studies have indeed shown a higher prevalence of heart failure in the Afro-Caribbean and Afro-American population with etiologies that differ from the Caucasian population. Among them, transthyretin (TTR) amyloidosis is rare in Europe but very common in African descendants with a prevalence of 3.4% of a transthyretin gene mutation (V122l) in this population (likely to induce hereditary amyloidosis after the fifth decade). It is a serious disease with a median survival of 2 to 6 years depending on the study and is often under-diagnosed with late detection at the time of a major cardiovascular event, such as a stroke or acute heart failure. Screening is done by imaging (cardiac MRI or bone scintigraphy with labelled diphosphonates). According to a study carried out in the Cardiology Department of the Martinique University Hospital (TEAM Amyloidosis study), one out of three left ventricular hypertrophy (LVH) (parietal thickness ≥ 15 mm), diagnosed by echocardiography, is amyloidosis. A study published by Thibaud Damy's team in 2015 already found a 5% prevalence of TTR gene mutation in patients with LVH. It is now accepted that systematic screening for amyloidosis is necessary in cases of LVH > 12 mm associated with at least one risk factor for amyloidosis ("red flags") in order to implement appropriate therapies and thus improve patient survival.

The study by Dungu et al. reports that cardiac amyloidosis is an underestimated etiology of acute heart failure in Afro-Caribbean immigrants in London. The study found a high prevalence of cardiac amyloidosis at 11.4% among 211 African-Caribbean immigrants compared to a Caucasian population (1.6%), with a higher mortality of these patients compared to patients with another cause of heart failure (median survival 2.3 years versus 7 years for other etiologies). The study by Arvanitis et al. describes a 5.1% prevalence of the transthyretin gene mutation (V122l) in 101 African Americans with heart failure (compared to 8.5% of mutation carriers among African-Caribbean immigrants in the Dungu study).

In these two studies, the prevalences of amyloidosis and the V122I mutation are probably underestimated, given the absence of systematic screening of all heart failure cases and the fact that only patients with left ventricular hypertrophy on transthoracic echography were targeted.

In addition, amyloidosis can take different forms from those usually described. Occasional observations in our experience at the University Hospital of Martinique have found cases of heart failure with dilated cardiomyopathy (DCM), associated with transthyretin cardiac amyloidosis. Several similar observations have been found in the literature.

The study hypothesise is that cardiac amyloidosis is as common, or more common, in acute heart failure in the French West Indies than elsewhere. A systematic screening for amyloidosis in all patients with acute heart failure would allow early initiation of appropriate treatment and improve their long-term outcome.

ELIGIBILITY:
Inclusion Criteria:

* Present functional or physical signs of acute heart failure (exertional dyspnea, orthopnea, paroxysmal nocturnal dyspnea, fatigue, jugular turgor, hepato-jugular reflux, edema of the lower limbs, galloping noise, crackles on pulmonary auscultation)
* BNP >100pg/mL or NT-proBNP >300pg/mL
* Diagnosis of heart failure confirmed by the cardiologist
* Be affiliated to a social security plan or beneficiary
* Be able to receive and understand information related to the research
* Able to freely express his/her non-opposition or informed and written consent.

Exclusion Criteria:

* Person under legal protection (guardianship, curatorship, safeguard of justice), and person deprived of liberty.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cardiac amyloidosis in acute heart failure patients in the French West Indies | 18 months +/- 8 days post inclusion
  The prevalence of cardiac amyloidosis in acute heart failure patients in Martinique and Guadeloupe over the study period will be determined by the following ratio
  Number of cardiac amyloidosis (old + new cases) in acute heart failure patients with hospital referral over the study period divided by the total number of acute heart failure patients with hospital referral over the period concerned
  This prevalence will be expressed per 10,000 and 100,000 people.

SECONDARY OUTCOMES:
Patient demographic characteristics | Baseline
  Age, gender, ethnicity, locality
To compare the clinical characteristics of heart failure patients with cardiac amyloidosis to other causes of heart failure | Baseline
  New York Heart Association (NYHA) stage, Heart failure picture
To compare the biological (total bilirubin) characteristics of heart failure patients with cardiac amyloidosis to other causes of heart failure | Baseline
  Biological assessment heart failure (total bilirubin) expressed in mg/L
To compare the biological (BNP or NT-proBNP) characteristics of heart failure patients with cardiac amyloidosis to other causes of heart failure | Baseline
  Biological assessment heart failure (BNP or NT-proBNP) expressed in pg/mL
To compare the biological (thyroid stimulating hormone) characteristics of heart failure patients with cardiac amyloidosis to other causes of heart failure | Baseline
  Biological assessment heart failure (thyroid stimulating hormone) expressed in mUI/l
To compare the biological (High-sensitivity (hs) cardiac troponin (cTn)) characteristics of heart failure patients with cardiac amyloidosis to other causes of heart failure | Baseline
  Biological assessment heart failure (High-sensitivity (hs) cardiac troponin (cTn)) expressed in µg/L
To compare the genotypic characteristics of heart failure patients with cardiac amyloidosis to other causes of heart failure | Baseline or through visit T2, an average of 6 months
  Presence of a mutation in the transthyretin gene
Describe the cases of amyloidosis identified according to the severity of cardiac involvement | Baseline
  Extra-cardiac impact (renal and liver function)
Describe the cases of amyloidosis according to the severity of the heart failure | Baseline
  Biomarkers (brain natriuretic peptide (BNP) or N-terminal fragment of probrain natriuretic peptide (NT-proBNP), High-sensitivity (hs) cardiac troponin (cTn)), etc expressed in sub-units of grams / sub-units of liters
Ultrasound criteria predictive of amyloid with or no LVH ≥12 mm | Baseline or up to 24 weeks post inclusion
  Ultrasound criteria predictive of amyloid involvement according to the presence or absence of LVH ≥12 mm by detailed analysis of cardiac echography
Diagnostic score for cardiac amyloidosis in acute heart failure | Through study completion, an average of 1 year
  This score will be composed of clinical, biological and imaging characteristics significantly associated with the presence of cardiac amyloidosis in a heart failure patient following the implementation of multivariate logistic regression modelling. The internal validation of this score will be determined by assessing :
  * The discrimination parameters of the score: sensitivity, specificity, and area under the Receiver Operating Characteristic (RO)C curve
  * Calibration of the score: comparison of predicted and observed risks (Hosmer-Lemeshow test).

CONTACTS AND LOCATIONS:
Overall Officials: Astrid MONFORT BRAFINE, MD, Study Director — CHU de Martinique
Locations (2):
- Laurent LARIFLA, Pointe-à-Pitre, Guadeloupe
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Result] Gabet A, Juilliere Y, Lamarche-Vadel A, Vernay M, Olie V. National trends in rate of patients hospitalized for heart failure and heart failure mortality in France, 2000-2012. Eur J Heart Fail. 2015 Jun;17(6):583-90. doi: 10.1002/ejhf.284. Epub 2015 May 6. PMID 25950872
- [Result] Dungu JN, Papadopoulou SA, Wykes K, Mahmood I, Marshall J, Valencia O, Fontana M, Whelan CJ, Gillmore JD, Hawkins PN, Anderson LJ. Afro-Caribbean Heart Failure in the United Kingdom: Cause, Outcomes, and ATTR V122I Cardiac Amyloidosis. Circ Heart Fail. 2016 Sep;9(9):e003352. doi: 10.1161/CIRCHEARTFAILURE.116.003352. PMID 27618855
- [Result] Arvanitis M, Chan GG, Jacobson DR, Berk JL, Connors LH, Ruberg FL. Prevalence of mutant ATTR cardiac amyloidosis in elderly African Americans with heart failure. Amyloid. 2017 Dec;24(4):253-255. doi: 10.1080/13506129.2017.1391086. Epub 2017 Oct 20. No abstract available. PMID 29052438
- See also: Frequency of cardiac amyloidosis inpatients with unexplained left ventricular hypertrophy: The Caribbean Amyloidosis Study — https://doi.org/10.1016/j.acvdsp.2017.11.055